CLINICAL TRIAL: NCT06714240
Title: Increased Protein Amount as a Nutritional Strategy to Enhance Muscle Protein Synthesis in ICU Patients
Brief Title: Enhanced Protein Intake to Support Muscle Protein Synthesis in ICU
Acronym: IPA-IC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2024/223
Record Dates: First submitted 2024-11-20; First posted 2024-12-03 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-10

CONDITIONS: Critical Illness; Muscle Protein Synthetic Response to Protein
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: The study is a prospective, randomized, longitudinal, controlled interventional trial with a parallel-group design.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal protein amount (Active Comparator)
  Interventions: Dietary Supplement: Nutritionally complete Tube Feed with standard protein levels
- Elevated protein amount (Experimental)
  Interventions: Dietary Supplement: Nutritionally complete Tube Feed with higher protein levels

INTERVENTIONS:
Dietary Supplement: Nutritionally complete Tube Feed with standard protein levels — Containing standard protein levels to target normal protein amount of 0.8 g of protein/kg body weight/day
  Arms: Normal protein amount
Dietary Supplement: Nutritionally complete Tube Feed with higher protein levels — Containing higher protein levels to target elevated protein amount of 1.3 g of protein/kg body weight/day.
  Arms: Elevated protein amount

SUMMARY:
Rationale - Critically ill patients often experience severe skeletal muscle wasting due to an imbalance between muscle protein synthesis (MPS) and degradation, contributing to long-term impairments such as ICU-acquired weakness (ICU-AW) and post-intensive care syndrome (PICS). Effective interventions to mitigate muscle wasting remain a critical unmet need. Protein intake has been identified as a potential modulator of MPS, but anabolic resistance and conflicting evidence regarding optimal protein intake necessitate further investigation.

Objective/Hypothesis - This study aims to evaluate the effect of a normal (target: 0.8 g protein/kg/day) versus elevated (target: 1.3 g protein/kg/day) protein intake on MPS rates over four days in critically ill patients.

Population - 26 critically ill patients who are suitable for enteral nutrition, mechanically ventilated (min 3 days), and stay at the ICU for at least 7 days will be included.

Method: Patients are randomly assigned to two groups (normal or higher protein intake). Muscle biopsies and blood samples will be collected to assess muscle protein synthesis rates.

DETAILED DESCRIPTION:
Complexities of Critical Illness - Critical illness encompasses the progression of severe medical conditions like major trauma or sepsis, which disrupt the body's homeostasis. This imbalance increases susceptibility to vital organ dysfunction, thereby posing imminent life-threatening consequences without prompt intensive medical support in hospitals. A key concern in critically ill patients is the rapid onset of skeletal muscle wasting, resulting in a condition known as intensive care unit-acquired weakness (ICU-AW). This muscle weakness is closely associated with extended mechanical ventilation and higher morbidity and mortality rates. Even after recovery, patients often suffer from long-term physical impairments and disabilities, resulting in post-intensive care syndrome (PICS), a condition characterized by persistent and debilitating consequences of ICU admission. Muscle weakness can last several years after ICU discharge, contributing to increased healthcare costs and a reduced quality of life. Considering the profound impact on both short- and long-term outcomes, coupled with the absence of effective strategies to prevent muscle wasting and weakness, remain major challenges in modern intensive care medicine.

Skeletal Muscle Protein Imbalance - Skeletal muscle mass is regulated by the balance between muscle protein synthesis, degradation, and folding. Under stable conditions, proteins serve structural and functional purposes crucial for growth, recovery, and adaptation. However, critical illness alters protein dynamics. Disturbance in protein folding can result in the accumulation of damaged proteins, causing a decline in protein quality, while imbalances between protein synthesis and degradation can lead to a decrease in quantity. Critically ill patients often experience a metabolic shift towards a catabolic state, wherein skeletal muscles are broken down to fulfill energy demands. Notably, during this catabolic phase, muscle proteins become a primary fuel source, with rates of muscle protein breakdown surpassing those of synthesis. This rapid muscle protein loss can result in up to 18% reduction in muscle mass within the first 10 days of ICU stay, ultimately leading to muscle atrophy.

Previous research has utilized nitrogen balance assessments and stable isotope techniques to evaluate whole-body protein turnover. However, only a few studies have specifically measured muscle protein synthesis (MPS) rates in critically ill patients using intravenous stable isotope infusions. These measurements typically cover short durations (less than 9 hours), making it challenging to extrapolate the findings to long-term outcomes due to the inherent limitations of amino acid tracer techniques. Adaptions to muscle disuse, inflammation, and catabolic stress likely occur over several days or weeks rather than hours. A promising alternative is oral deuterated water (D2O), which enables the assessment of MPS over longer periods (days or weeks). Current research by our group used D2O to provide insights into muscle synthesis rates over multiple ICU days. This pioneering study will establish critical baseline data for future research.

Protein Ingestion as a Key Modulator - To improve patient recovery, interventions targeting muscle loss are recommended. The 2019 guidelines from the European Society for Clinical Nutrition and Metabolism (ESPEN) emphasize the importance of nutritional support for mechanically ventilated ICU patients. Specifically, dietary proteins and their amino acid composition are key in mitigating skeletal muscle wasting and improving long-term clinical outcomes. However, the efficacy of dietary protein to stimulate MPS is regulated by various physiological factors such as dietary protein digestion and amino acid absorption, splanchnic amino acid retention, postprandial insulin release, skeletal muscle tissue perfusion, amino acid uptake by muscle, and intramyocellular signaling. Current international guidelines recommend elevated protein intake for critically ill patients, ranging from 1.2 to 2.0 g protein/kg body weight/day, exceeding recommendations for healthy individuals. However, while higher protein intake has been shown to enhance MPS, recent research suggests that the upper threshold of 2.0 g/kg/day may negatively impact health-related quality of life without improving functional outcomes up to 180 days post-ICU admission. Given these conflicting findings, the precise impact of elevated protein intake on MPS in critically ill patients remains unclear, warranting further investigation to determine the optimal protein requirements during critical illness. Furthermore, despite these widely accepted guidelines and intake recommendations, observational studies have reported that actual protein intake in ICU patients often falls below these targets, ranging from 0.7 to 1.2 g/kg/day. Recent research demonstrated efficient digestion and absorption of enterally administered protein. Nevertheless, post-prandial muscle protein synthesis rates were much lower in critically ill patients than in healthy volunteers. This indicates that critical illness does not impair dietary protein digestion and amino acid absorption. However, incorporating dietary protein-derived amino acids into skeletal muscle protein is blunted, representing anabolic resistance to dietary protein. This anabolic resistance underscores the complexity of muscle protein metabolism in critically ill patients and highlights the need for effective strategies to attenuate skeletal muscle wasting.

In short, this prospective study aims to evaluate the effect of normal vs. elevated enteral protein administration on muscle protein synthesis rates and muscle characteristics in critically ill patients. This research will provide valuable insights to develop effective nutritional interventions to address skeletal muscle wasting in critical illness.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Suitability for enteral nutrition (i.e., no GI failure, absence of complete intestinal obstruction, no major intra-abdominal sepsis)
* Expected mechanical ventilation of minimal three days
* Expected ICU stay of at least seven days

Exclusion Criteria:

* BMI ≥ 40 kg/m²
* Spinal cord injury
* Chronic corticosteroid use before hospital admission
* severe allergies or intolerances (e.g., to cow's milk protein, fish, soy, pea protein or galactosemia)
* Severe kidney and/or liver failure
* Requirements for dialysis
* Bleeding disorders, including anticoagulant and antiplatelet therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Myofibrillar protein fractional synthetic rate | 1-4 days
  The myofibrillar protein synthesis rates are calculated using D2O.

SECONDARY OUTCOMES:
Mixed muscle protein fractional synthetic rate | 1-4 days
  The mixed muscle protein synthesis rates are calculated using D2O.
Plasma amino acids concentrations | 1-4 days
  Determining differences in plasma amino acids concentration between groups receiving normal versus elevated protein levels through enteral nutrition
Muscle fiber size in µm² | Final intervention day (after 4 days of enteral feeding)
  Muscle fiber size will be assessed using immunofluorescence staining.
Proportion (%) of muscle fiber types (type I and type II) | Final intervention day (after 4 days of enteral feeding)
  Fiber proportion will be assessed using immunofluorescence staining.
Myonuclei quantity | Final intervention day (after 4 days of enteral feeding)
  Myonuclei quantity will be assessed using immunofluorescence staining.
Mitochondrial respiration | Final intervention day (after 4 days of enteral feeding)
  Mitochondrial respiration will be assessed using Oroboros Instruments (Oroboros O2k FluoRepirometer).

OTHER OUTCOMES:
Age in years | Baseline
  Heteroanamnesia
Body mass in kg | Baseline
  Heteroanamnesia
Height in m | Baseline
  Heteroanamnesia
BMI in kg/m² | Baseline
  Calculated from height and body mass
Clinical health data | Baseline
  Clinical health data (Smoker status, Reason for ICU admission, Comorbidities, Highest recorded temperature, Respiratory rate, Blood pressure, Heart rate, Glasgow Coma Scale, Charlson Comorbidity Index, Rockwood Clinical Frailty Index, APACHE II score, APACHE IV score, APS score, SAPS II, Medications, Routine blood test results, Length of ICU and hospital stay, Days in study, Survival outcomes, Muscle biopsy time points, Nutritional intake, Study product compliance, Study product tolerance) will be collected by the attending physician, healthcare staff, and the laboratory technicians.

CONTACTS AND LOCATIONS:
Locations (1):
- Jessa Hospital Campus Virga Jesse, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No